CLINICAL TRIAL: NCT07071311
Title: Using a Mobile Health (mHealth) Self-Guided Application in the Workplace
Brief Title: Can Mindsets Predict Help-Seeking? A Growth Mindset Intervention and Mental Health App Engagement in Working Adults
Acronym: GROW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intellect Pte. Ltd. (Industry)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NUS-IRB-2022-253
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: App Engagement; Employee Health; Mobile Apps; Self-care Tools; Mindsets
Keywords: App Engagement; Behavior Change; Growth Mindset; Mobile App; mHealth; Self-help; Self-care; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This single-session growth mindset intervention consists of reading and reflective writing activities that present mental health as something that can be improved, rather than something fixed. The goal is to show that adopting a growth mindset of mental health can encourage more proactive mental health behaviors.
  To begin, participants read stories of three employees who share their personal experiences navigating mental health challenges in the workplace. Each story highlights the employee's struggles, how they came to see mental health as changeable, and the steps they took to care for their well-being (e.g., practicing self-care or seeking therapy). After reading, participants complete a short reflective essay in response to three prompts. These prompts guide them to examine their own mindset about mental health, endorse a growth mindset towards mental health, and outline specific actions they can take to proactively support their own mental well-being.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Technology Condition (Placebo Comparator): This single-session control exercise aims to encourage the use of digital technology in the workplace. It positions participants as experts who provide guidance to others on how to use digital tools more effectively at work.
  First, participants will read stories about employees' experiences navigating their workload with the help of workplace technology. Each story highlights the employee's initial struggles with learning new digital tools and how they eventually recognized the value of these technologies. This includes examples of how they viewed digital learning as manageable and took proactive steps-such as seeking help from colleagues or setting aside time to practice. Then, participants will complete a short reflective essay in response to three writing prompts. These prompts guide them to reflect on their own experiences with digital tools and offer practical advice to others on how to use new technologies effectively in the workplace.
  Interventions: Behavioral: Digital Technology Condition
- Growth Mindset Intervention (Experimental): This single-session growth mindset intervention consists of reading and reflective writing activities that present mental health as something that can be improved, rather than something fixed. The goal is to show that adopting a growth mindset of mental health can encourage more proactive mental health behaviors.
  To begin, participants will read stories of three employees who share their personal experiences navigating mental health challenges in the workplace. Each story highlights the employee's struggles, how they came to see mental health as changeable, and the steps they took to care for their well-being (e.g., practicing self-care or seeking therapy). After reading, participants will complete a short reflective essay in response to three prompts. These prompts guide them to examine their own mindset about mental health, endorse a growth mindset towards mental health, and outline specific actions they can take to proactively support their own mental well-being.
  Interventions: Behavioral: Growth Mindset Intervention

INTERVENTIONS:
Behavioral: Growth Mindset Intervention — This single-session growth mindset intervention consists of reading and reflective writing activities that present mental health as something that can be improved, rather than something fixed. The goal is to show that adopting a growth mindset of mental health can encourage more proactive mental health behaviors.
  To begin, participants will read stories of three employees who share their personal experiences navigating mental health challenges in the workplace. Each story highlights the employee's struggles, how they came to see mental health as changeable, and the steps they took to care for their well-being (e.g., practicing self-care or seeking therapy). After reading, participants will complete a short reflective essay in response to three prompts. These prompts guide them to examine their own mindset about mental health, endorse a growth mindset towards mental health, and outline specific actions they can take to proactively support their own mental well-being.
  Arms: Growth Mindset Intervention
Behavioral: Digital Technology Condition — This single-session control exercise aims to encourage the use of digital technology in the workplace. It positions participants as experts who provide guidance to others on how to use digital tools more effectively at work.
  First, participants will read stories about employees' experiences navigating their workload with the help of workplace technology. Each story highlights the employee's initial struggles with learning new digital tools and how they eventually recognized the value of these technologies. This includes examples of how they viewed digital learning as manageable and took proactive steps-such as seeking help from colleagues or setting aside time to practice. Then, participants will complete a short reflective essay in response to three writing prompts. These prompts guide them to reflect on their own experiences with digital tools and offer practical advice to others on how to use new technologies effectively in the workplace.
  Arms: Digital Technology Condition

SUMMARY:
Despite the growing adoption of digital mental health initiatives in the workplace, employees' sustained engagement with these resources remained relatively low. Encouraging a growth mindset about mental health may help motivate employees to actively use these tools to support their well-being.

This randomized controlled trial (RCT) examines whether introducing a growth mindset intervention prior to using a mental health app can improve users' repeated engagement with the app.

ELIGIBILITY:
Inclusion Criteria:

* Being able to read and understand English
* Being 18 years or older
* Being employed
* Not using other mental health mobile applications or services concurrently.

Exclusion Criteria:

* Not able to read and understand English
* Younger than 18 years old
* Unemployed
* Using other mental health mobile applications or services concurrently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Repeated App Engagement | Repeated Engagement was defined as whether participants completed more than one self-help feature within three months of the growth mindset intervention
  Completion of >1 self-guided feature on the mental health app ("Intellect")

SECONDARY OUTCOMES:
Anxiety and Depressive Symptoms | Baseline Assessment
  Participants' baseline anxiety and depressive symptoms were assessed with the 4-item Patient Health Questionnaire. Scores are summed, ranging from 0-12. Higher PHQ-4 scores indicate more severe anxiety and depressive symptoms. The cutoffs for mild, moderate, and severe depression were 3, 6, and 9 respectively.
Perceived Stress | Baseline Assessment
  Participants' baseline stress levels over the last month were assessed using the 4-item Perceived Stress Scale. Scores are summed, ranging from 4-20, with higher scores indicating greater perceived stress.
Positive Well-being | Baseline Assessment
  Participants' baseline positive well-being was assessed using the 7-item Short Warwick-Edinburgh Mental Wellbeing Scale. Scores are summed, ranging from 7-35, with higher scores indicating more positive well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Intellect Pte Ltd., Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlies results in the publication
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 1 year after the publication of results

REFERENCES:
- [Background] Walton, G. M. (2014). The new science of wise psychological interventions. Current Directions in Psychological Science, 23(1), 73-82.